CLINICAL TRIAL: NCT03405675
Title: Gerontology Research Programme: Biological, Clinical, Psychosocial and Behavioural Predictors of Health Status in Prospectively Followed-up Cohorts of Elderly Persons
Brief Title: Gerontology Research Programme: The Singapore Longitudinal Ageing Studies (SLAS I & II)
Acronym: SLAS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Karolinska Institutet (Other); Tan Tock Seng Hospital (Other); Ng Teng Fong General Hospital (Other); St Luke's Hospital, Singapore (Other); St. Paul's Hospital, Canada (Other); Singapore Institute of Technology (Other); Duke-NUS Graduate Medical School (Other); Melbourne Health (Other); University of California (Other); University Hospital, Basel, Switzerland (Other); Université de Sherbrooke (Other); University Hospital Tuebingen (Other); National University Hospital, Singapore (Other); Khoo Teck Puat Hospital (Other); Shanghai Jiao Tong University School of Medicine (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, A/Prof Ng Tze Pin, Associate Professorial Fellow and Research Director, National University of Singapore
Other Study IDs: NUS-IRB 04-140
Record Dates: First submitted 2017-10-26; First posted 2018-01-23 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Cognitive Changes Due to Organic Disorder (Finding); Dementia; Mild Cognitive Impairment; Frailty; Depression; Healthy Ageing; Biological Ageing
Keywords: Dementia; Mild cognitive impairment; Cognitive abilities and changes; Functional change and disabilities; Depression; Health and social services utilization; Quality of life; Adverse drug effects; Social network and support; Self-rated health; Medical morbidities; Falls; Health risk behaviors; Nutrition; Apo-E lipoprotein; Phytochemicals; B12; Folate; Homocysteine; Lifestyle; Physical activity; Leisure activity; Successful ageing; Mortality
MeSH Terms: conditions — Signs and Symptoms; Dementia; Cognitive Dysfunction; Frailty; Depression; Drug-Related Side Effects and Adverse Reactions; Health Risk Behaviors; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological specimens (blood and urine) will be analyzed for full blood count, lipid panel, liver function test, blood biochemistry, PBMC, DNA, immunological tests (whole blood, serum, plasma).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SLAS 1: The subjects (N=2800) are recruited from all residents aged 55 years and above in Singapore in the areas covered by the South-East Community Development Council: Geylang, Aljunied, MacPherson, Marine Parade and Bedok (SLAS-I).
  Interventions: Other: SLAS 1
- SLAS 2: An additional 3200 subjects are recruited from residents in the Bukit Merah and Jurong (SLAS-II).
  Interventions: Other: SLAS 2

INTERVENTIONS:
Other: SLAS 1 — NA. Observational study, no interventions administered.
  Groups: SLAS 1
Other: SLAS 2 — NA. Observational study, no interventions administered.
  Groups: SLAS 2

SUMMARY:
The Gerontology Research Programme (GRP) in the National University Singapore's Department of Psychological Medicine, was formed to coordinate and facilitate the conduct of multi-disciplinary research on in a wide range of research on ageing and health. The establishment of the Singapore Longitudinal Aging Cohort will provide a large community-based cohort of elderly subjects for observational studies with useful clinical applications. Research synergy is achieved in terms of pooling multi-disciplinary expertise, and combining genetic, biological, environmental, behavioural, social, clinical, and health services approaches to gerontological research.

DETAILED DESCRIPTION:
The SLAS is the principal longitudinal cohort study in GRP. The SLAS is a community-based longitudinal epidemiologic study that aims to increase the understanding of ageing and health, and the factors that influence the ageing process. SLAS seeks to identify the cognitive, biomedical, lifestyle and behavioral, as well as psychosocial risk and protective factors that affect the transition from healthy ageing to functional impairment, illness and death.

Participants recruited into SLAS are community-dwelling seniors, aged 55 and above, from various areas in Singapore. Participants are approached door-to-door, are provided detailed information regarding their participation, and are required to provide informed consent before enrollment into the study. The study procedure includes a baseline survey upon enrollment, and participants are revisited on a 3-yearly basis thereafter.

Enrolled subjects provide baseline data through structured interviews, physician assessments, laboratory testing, and self-reports of conditions, symptoms, and risk behaviors. Data in the study is collected by trained research staff and nurses. The information to be collected include:

Outcomes:

Primary Outcomes

4 Main Primary Outcomes

1. Mild cognitive impairment and cognitive functioning
2. Frailty
3. Depression, anxiety (Mood disorder I)
4. Successful and healthy ageing

Basic screening followed by diagnostic tests.

Cognitive domain functioning. Particpants are screened fro cogntve impairment using global cognitive tests (MMSE and MOCA). An exhaustive neuropsychological assessment battery is also conducted to assess specific cognitive domain functioning of participants. Selected participants that meet screening criteria, thus indicating the presence of possible cognitive impairment, undergo further testing to determine their cognitive functioning status (cognitively normal, mild cognitive impairment, cognitive decline, or dementia), as diagnosed by a panel of geriatricians, in accordance with the DSM-IV-TR criteria for dementia (1), and the MCI Working Group of the European Consortium on Alzheimer's disease criteria (2).

Frailty assessment. A battery of measures, including self-report, physical assessments and anthropometric measures, is administered to measure the frailty status of the individuals, in accordance with the Fried et al.'s phenotype criteria (3).

Psychiatric assessment. Several self-reported questionnaires are administered to measure the symptomatology of common psychiatric disorders such as depression, among others. Selected participants that meet screening criteria, thus indicating the presence of possible psychiatric disorders, would undergo further testing to determine their mental health state, in accordance with the DSM-IV-TR criteria (1).

Successful and healthy ageing. Successful and healthy ageing is determined by a number of self-reported and objective measurements of health which aim to reflect the overall and physical health, cognitive, emotional and social well-functioning (inclusive of life engagement and life satisfaction) of the individual.

Secondary Outcomes

Physical domain functioning. Self-reported measures as well as physical assessments would be conducted to measure physical functioning, disability and independence in activities of daily living among participants.

Health, health services utilization. Data regarding the history of chronic medical conditions and falls, medication use, use of hospital and primary care services and self-rated health.

Quality of Life. Self-reported measures would be conducted to measure the quality of life amongst the participants.

Mortality. The date of death of participants would be recorded, as well as assessing the Singapore National Registry of Diseases Office (NRDO).

Respiratory functioning. Data regarding respiratory functioning would be collected via a spirometry test.

Risk and protective factors:

Socioeconomic and demographic variables. Information regarding the age, gender, educational status and household income would be collected from the participants via self-report.

Medical history. Information regarding the history of selected medical and mental disorders would be collected from the participants via self-report.

Biological determinants. Biological specimens (blood and urine) will be analyzed for constituents of interest (e.g. micronutrients, lipid and glucose levels, among others).

Pharmacological determinants. The use of pharmacological agents such as anti-inflammatory, cholesterol-lowering and other drugs will be recorded via a self-report measure.

Nutrition. Participants would be assessed on their nutritional status and dietary consumption (NSI screening, MNA screening, food frequency, 2-day food diary). The dietary records are analyzed for nutrients of interest and phytochemicals such as B12, B6, folate, curcumin, and other nutritional supplements.

Lifestyle and health risk behaviors. Lifestyle behaviors measured would include physical, leisure and social activities engagement duration and frequency. Health risk behaviors measured include the body mass index and other anthropometric measures, smoking, customary physical activity, social and productive activities and alcohol use among participants.

Psycho-social data. Self-reported questionnaires are administered to measure life satisfaction, personality, religiosity, social support and asocial network connections for select participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to self-ambulate
* Adequate cognitive capacity for participation

Exclusion Criteria:

- Individuals with severe physical or mental disabilities were excluded.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-dwelling Elderly (>55 years old) that are able to self-ambulate and who possess sufficient cognitive capacity for participation. Individuals with severe physical or mental disabilities were excluded.
Sampling Method: Probability Sample
Enrollment: 6183 (Actual)
Dates: Start 2003-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Dementia and Mild Cognitive Impairment (MCI) Subtyping (Clinical diagnosis of different stages of Dementia) | 20 years - once every 3-4 years
  Dementia and MCI is determined by clinical case conference adjudication where geriatric and psychiatric clinicians convene to determine the diagnosis of a case, utilizing the data from (i) Mini Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA) (4-5); (ii) Clinical Dementia rating scale: a 5-point scale used to characterize 6 cognitive and functional domain performance: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care (6). Information to make each rating is obtained through a semi-structured interview of the patient and a reliable informant (e.g. family member). A higher score indicates increased severity of cognitive impairment; (iii) Informant Questionnaire of Cognitive Decline in the Elderly (IQCODE) - reliable informants report on the cognitive state of the participant (7); (iv) a scale on self-reported subjective cognitive difficulties; and (v) a neuropsychological assessment battery (described below).
Global and specific domain cognitive functioning ability (Measuring of Global and Specific domain of Cognitive functions) | 20 years - once every 3-4 years
  MMSE (4) and MoCA (5) - 30 items, total scores range from 0-30, higher scores indicate better cognitive functioning. A cut-off of a score of =<25 is determined as screening positive for cognitive impairment.
  Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) (8) - measures immediate memory, visuospatial ability, language, attention, delayed memory, and a global cognitive functioning score (a summation of domain scores).
  A neurocognitive battery measures immediate and delayed memory/learning, visuospatial ability, language, attention, and executive functioning. All domains are calculated by weighted averages of age and education adjusted scores. Tests: (i) Digit Span forward and backwards tasks (9); (ii) Rey's Auditory Verbal Learning Test (10); (iii) Story Memory Test (11); (iv) Brief Visuospatial Memory Test - Revised (12); (v) Boston Naming Test (13); (vi) Clock Reading Test; (viii) Colour Trials 1 and 2 (14); (ix) Block Design task (9).
Frailty (Measuring the physical and Cognitive Frailty) | 20 years - once every 3-4 years
  Physical frailty was assessed by scores (1 = present, 0 = absent) for five components (shrinking, weakness, slowness, exhaustion, and low Physical Activity (PA)) proposed by Fried et al (3), with the following operational modifications: (i) Shrinking was defined by unintentional weight loss of 4 kg or more in the past 6 months, or BMI less than 18.5 kg/m2, or calf circumference of 31 cm or less. (ii) Weakness was assessed by knee extension strength task in kilogram. (iii) Slowness was assessed by a gait speed test (15). (iv) Exhaustion was measured as a summed score of 3 questions (1-5), "Did you have lots of energy/feel tired (reverse-scored, rs)/worn out (rs)?" (16). A score of <10 was used to denote exhaustion. (v) Low PA was measured by the LASA PA scale, with those falling below the local gender-specific lowest quintile deemed as low PA (17). Participants are categorised by their total scores as robust (score = 0), pre-frail (score = 1-2), and frail (score = 3-5).
Depressive symptoms and diagnosis (Measuring of Depressive symptoms and assessment of stages of Depression) | 20 years - once every 3-4 years
  Depressive symptoms are assessed by the 15-item version of the Geriatric Depression Scale (GDS), with a higher score indicating higher depressivity (18). A cut-off score of 5 is used as indicating the presence of depression. Additionally, participants are formally diagnosed by a medically trained research fellow for common mood-related psychiatric conditions using the Structured Clinical Interview for DSM Disorders (SCID) of DSM IV-TR (1), such as Major Depressive Disorder, Minor Depression, Dysthmic Disorder, Mania/Hypomania disorder, Anxiety and panic disorder, Obsessive-compulsive disorder, Post traumatic stress disorder, Psychotic disorder, Mood disorder due to a General Medical Condition and Alcohol abuse disorders, if they screen as positive for depression on the GDS.
Successful ageing (Measuring the biological, psycho-social and lifestyle factors associated with Successful Ageing) | 20 years - once every 3-4 years
  Successful aging is previously defined (25). Briefly, a score of successful ageing reflects the overall and physical health, cognitive, emotional, social well-functioning, including life engagement & satisfaction. Physical health and functional well-being was defined as a "good/excellent" self-reported health and IADL independence (20). Cognitive well-functioning and emotional wellbeing was denoted by a minimum MMSE score of 26 (4), and a score below 5 on the GDS (≤5) (18). Social functioning and active engagement in life activities was assessed using a validated questionnaire (26) on participation levels in social, recreational, civic activities, voluntary work, employment/business, and domestic activities. Overall positive life satisfaction was determined using the Life Satisfaction Scale that assessed interest in life, happiness, loneliness, and general ease of living (27). Total summed score ranges from 4 to 18, with the lowest decile indicating a positive life satisfaction.

SECONDARY OUTCOMES:
Self-reported independent functioning (Measuring the BADL and IADL) | 20 years - once every 3-4 years
  Self-reported Independent Functioning is assessed using the Barthel Index (19) and the Lawton and Brody Instrumental Activity of Daily Living Inventory (20), whereby participants report the degree of dependence on others for several daily and instrumental tasks.
Physical performance (Measuring the physical performance tests) | 20 years - once every 3-4 years
  Assessed by the Physical Performance Battery which includes the Performance-Oriented Mobility Assessment-Balance and Gait scales (21-22), with a higher score indicating a higher performance in terms of balance or gait; as well as the amount of force displaced in Newtons on a handgrip and knee extension dynamometer. The scores for each of the tests would be combined into a weighted average that reflects overall physical performance.
Health services utilization (Measuring cost and frequency of health services utilization) | 20 years - once every 3-4 years
  Self-reported frequency of doctor visits over a past 12-month period.
Quality of life (Measuring the Quality of life SF 12) | 20 years - once every 3-4 years
  Assessed by self-reported scales: (i) EQ5D- 3L - a measure of health-related quality of life that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale (23). (ii) 12-Item Short Form Survey (SF-12) is a 12-item questionnaire used to assess generic health outcomes from the patient's perspective, covering the eight domains of health outcomes: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional & mental health (24).
Mortality (Measuring the risk factors related to mortality) | 20 years
  Date and cause of death data is collected by computerized record linkage with the National Death Registry through the Singapore National Registry of Diseases Office (NRDO).
Post-bronchodilation spirometry (Measuring the lung functions tests) | 20 years - once every 3-4 years
  A measurement of lung function which yields the (i) Forced vital capacity - the determination of the vital capacity from a maximally forced expiratory effort; (ii) the FEV1 - volume that has been exhaled at the end of the first second of forced expiration; and the (iii) Peak expiratory flow: The highest forced expiratory flow measured with a peak flow meter. Measurements are made following American Thoracic Society (ATS) criteria for spirometric standardization and procedures, based on the best of four readings, with less than 5% variation in the two best readings. FEV1 is expressed as the percentage of predicted from local norms.

CONTACTS AND LOCATIONS:
Overall Officials: Tze Pin Ng, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and statistical manual of Mental Disorders, (4th ed., text rev.; DSM-IV-TR). American Psychiatric Association, Washington. 2000.
- [Background] Portet F, Ousset PJ, Visser PJ, Frisoni GB, Nobili F, Scheltens P, Vellas B, Touchon J; MCI Working Group of the European Consortium on Alzheimer's Disease (EADC). Mild cognitive impairment (MCI) in medical practice: a critical review of the concept and new diagnostic procedure. Report of the MCI Working Group of the European Consortium on Alzheimer's Disease. J Neurol Neurosurg Psychiatry. 2006 Jun;77(6):714-8. doi: 10.1136/jnnp.2005.085332. Epub 2006 Mar 20. PMID 16549412
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Folstein MF, Folstein SE, McHugh PR, Fanjiang G. Mini-Mental State Examination: MMSE user's guide. Psychology Assessment Resources; 2000.
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] O'Bryant SE, Waring SC, Cullum CM, Hall J, Lacritz L, Massman PJ, Lupo PJ, Reisch JS, Doody R; Texas Alzheimer's Research Consortium. Staging dementia using Clinical Dementia Rating Scale Sum of Boxes scores: a Texas Alzheimer's research consortium study. Arch Neurol. 2008 Aug;65(8):1091-5. doi: 10.1001/archneur.65.8.1091. PMID 18695059
- [Background] Jorm AF. A short form of the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE): development and cross-validation. Psychol Med. 1994 Feb;24(1):145-53. doi: 10.1017/s003329170002691x. PMID 8208879
- [Background] Randolph C, Tierney MC, Mohr E, Chase TN. The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity. J Clin Exp Neuropsychol. 1998 Jun;20(3):310-9. doi: 10.1076/jcen.20.3.310.823. PMID 9845158
- [Background] Wechsler D. Wechsler adult intelligence scale-fourth. San Antonio, TX: The Psychological Corporation Google Scholar; 2008.
- [Background] Rey A. L'examen psychologique dans les cas d'encéphalopathie traumatique.(Les problems.). Archives de psychologie (1941).
- [Background] Yeo D, Gabriel C, Chen C, Lee S, Loenneker T, Wong M. Pilot validation of a customized neuropsychological battery in elderly Singaporeans. Neurol J South East Asia 1997 2(123).
- [Background] Benedict RHB. Brief visuospatial memory test - revised: Professional manual. Lutz, FL: Psychological Assessment Resources, Inc; 1997.
- [Background] Kaplan E, Goodglass H, Weintraub S. Boston naming test. Pro-ed; 2001.
- [Background] D'Elia LF, Satz P, Uchiyama CL, White T. Color Trails Test: Professional Manual. Odessa (Florida): Psychological Assessment Resources; 1996.
- [Background] Kluger A, Gianutsos JG, Golomb J, Wagner A Jr, Wagner D, Scheurich S. Clinical features of MCI: motor changes. Int Psychogeriatr. 2008 Feb;20(1):32-9. doi: 10.1017/S1041610207006461. PMID 18072982
- [Background] Ware JE, Keller SD, Kosinski M. SF-12: How to Score the SF-12 Physical and Mental Health Summary Scales. Lincoln, RI: QualityMetric; 1998.
- [Background] Siebeling L, Wiebers S, Beem L, Puhan MA, Ter Riet G. Validity and reproducibility of a physical activity questionnaire for older adults: questionnaire versus accelerometer for assessing physical activity in older adults. Clin Epidemiol. 2012;4:171-80. doi: 10.2147/CLEP.S30848. Epub 2012 Jul 16. PMID 22866018
- [Background] Vinkers DJ, Gussekloo J, Stek ML, Westendorp RG, Van Der Mast RC. The 15-item Geriatric Depression Scale (GDS-15) detects changes in depressive symptoms after a major negative life event. The Leiden 85-plus Study. Int J Geriatr Psychiatry. 2004 Jan;19(1):80-4. doi: 10.1002/gps.1043. PMID 14716703
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Tinetti ME, Williams TF, Mayewski R. Fall risk index for elderly patients based on number of chronic disabilities. Am J Med. 1986 Mar;80(3):429-34. doi: 10.1016/0002-9343(86)90717-5. PMID 3953620
- [Background] Tinetti ME. Performance-oriented assessment of mobility problems in elderly patients. J Am Geriatr Soc. 1986 Feb;34(2):119-26. doi: 10.1111/j.1532-5415.1986.tb05480.x. No abstract available. PMID 3944402
- [Background] Rabin R, Oemar M, Oppe M, Janssen B, Herdman M. EQ-5D-3L User Guide: Basic information on how to use the EQ-5D-3L instrument. Rotterdam: EuroQol Group; 2011.
- [Background] Ware JE, Kolinski M, Keller SD. How to Score the SF-12 Physical and Mental Health Summaries: A User's Manual. Boston: The Health Institute, New England Medical Centre, Boston, MA; 1995.
- [Background] Ng TP, Broekman BF, Niti M, Gwee X, Kua EH. Determinants of successful aging using a multidimensional definition among Chinese elderly in Singapore. Am J Geriatr Psychiatry. 2009 May;17(5):407-16. doi: 10.1097/JGP.0b013e31819a808e. PMID 19390298
- [Background] Niti M, Yap KB, Kua EH, Tan CH, Ng TP. Physical, social and productive leisure activities, cognitive decline and interaction with APOE-epsilon 4 genotype in Chinese older adults. Int Psychogeriatr. 2008 Apr;20(2):237-51. doi: 10.1017/S1041610207006655. Epub 2008 Jan 11. PMID 18190728
- [Background] Koivumaa-Honkanen H, Honkanen R, Viinamaki H, Heikkila K, Kaprio J, Koskenvuo M. Self-reported life satisfaction and 20-year mortality in healthy Finnish adults. Am J Epidemiol. 2000 Nov 15;152(10):983-91. doi: 10.1093/aje/152.10.983. PMID 11092440
- [Derived] Ng TP, Lee TS, Lim WS, Chong MS, Yap P, Cheong CY, Rawtaer I, Liew TM, Gwee X, Gao Q, Yap KB. Functional mobility decline and incident mild cognitive impairment and early dementia in community-dwelling older adults: the Singapore Longitudinal Ageing Study. Age Ageing. 2022 Sep 2;51(9):afac182. doi: 10.1093/ageing/afac182. PMID 36074716